CLINICAL TRIAL: NCT03893149
Title: A Before-school Physical Activity Intervention Program to Improve Attention in Vulnerable Children: The Active-Start Trial
Brief Title: Attention Capacity and Before-school Physical Activity Intervention Program
Acronym: Active-Star
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N°: 938 USACH
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Physical Activity; Behavior; Child Behavior; Attention Deficit Hyperactivity Disorder
Keywords: Exercise; Prevention; Attention capacity
MeSH Terms: conditions — Motor Activity; Behavior; Child Behavior; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Start intervention (Experimental): Supervised exercise training
  Interventions: Behavioral: Active-Start intervention; Behavioral: No Intervention
- Control group (No Intervention): No-exercise

INTERVENTIONS:
Behavioral: Active-Start intervention — Supervised exercise training. The intervention is a physical activity intervention that consist of 5 times per week before starting the first school-class (8:00-8:30 a.m.), 5 times per week. Each session was previously planned and described in a manual dedicated to the study. These sessions were designed by the research team and delivered by a graduate in Sport The intervention program included sports games adapted to the age of the participants, playground games, dance and other recreational activities. The intensity of the main part of the sessions was moderate-to-vigorous according to a previous study and this intensity was confirmed by accelerometry. Also, different activities favoring social interactions were designed to facilitate the interactions between the participants at the end of the sessions (cold-down).
  Arms: Active-Start intervention
Behavioral: No Intervention — No-exercise
  Arms: Active-Start intervention

SUMMARY:
Despite the evidence and the potential of physical activity related to cognition and academic performance in children, the effects of a before-school physical activity program on these parameters remains unknown.

DETAILED DESCRIPTION:
Despite public health concerns and the extensively documented health benefits of physical activity, a large proportion of Chilean children do not meet the physical activity recommendations (Aguilar-Farias et al., 2018). Since most children spend a majority of their waking hours at school, this environment is appropriate for the implementation of preventive interventions, particularly those that include activities promoting physical activity (Naylor & McKay, 2009). With the absence of opportunities for physical activity during the school day, before-school programs have become a popular option to help children increasing their physical activity levels (Stylianou, van der Mars, et al., 2016). Although several recent studies support a positive effect of before school-based physical activity on health (Westcott, Puhala, Colligan, Loud, & Cobbett, 2015), less literature has evaluate the cognitive outcomes (Stylianou, Kulinna, et al., 2016) such as attention capacity.

ELIGIBILITY:
Inclusion Criteria:

* All students in fourth grade (aged 8-10 years)
* Children's parents/caregivers will give their written consent to the children's participation.
* Collaboration in the family to respond to questionnaires

Exclusion Criteria:

* Children with some physical pathology or medical contraindication to perform physical exercise
* Diagnosed with learning disabilities or mental disorders

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Selective attention | Change from Baseline and 8-weeks immediately after the interventions ends
  The D2- Test were used as indicators of selective attention

SECONDARY OUTCOMES:
Academic performance | Change from Baseline and 8-weeks immediately after the interventions ends
  Was recorded by 2018-2019 year final exam scores
Executive function | Change from Baseline and 8-weeks immediately after the interventions ends
  The D2- Test were used as indicators of cognitive flexibility
Body fat percentage | Change from Baseline and 8-weeks immediately after the interventions ends
  Was recorded by bioelectrical impedance analysis
Body mass index | Change from Baseline and 8-weeks immediately after the interventions ends
  Weight and height were used to calculate BMI (weight in kilograms divided by the square of height in meters).
Waist circumference | Change from Baseline and 8-weeks immediately after the interventions ends
  Waist circumference was measured in the horizontal plane at the superior border of the right iliac crest.
Fat free mass | Change from Baseline and 8-weeks immediately after the interventions ends
  Was recorded by bioelectrical impedance analysis
Muscular strength | Change from Baseline and 8-weeks immediately after the interventions ends
  The handgrip test, each child performed the test twice with each hand, and the maximum value of each hand was taken and averaged
Standing long jump test | Change from Baseline and 8-weeks immediately after the interventions ends
  The longest attempt from 3 was recorded (centimeters) and multiplied by the body weight to obtain an absolute measurement
4x10-m shuttle-run test | Change from Baseline and 8-weeks immediately after the interventions ends
  The speed-agility was assessed twice using the 4 x 10-m shuttle-run test and the fastest completion time (seconds) was recorded
Cardiorespiratory fitness | Change from Baseline and 8-weeks immediately after the interventions ends
  Cardiorespiratory fitness was assessed through the 20-m shuttle-run test and the total number of completed laps was registered
Blood pressure | Change from Baseline and 8-weeks immediately after the interventions ends
  Blood pressure was recorded by a automatic sphygmomanometer with the arm supported at heart level after sitting quietly for 10 min
Mediterranean diet | Change from Baseline and 8-weeks immediately after the interventions ends
  This information was self-reported by the children withguided assistance by a trained psychologis with Mediterranean diet (Kidmed) tool

CONTACTS AND LOCATIONS:
Overall Officials: Antonio García-Hermoso, PhD, Principal Investigator — Universidad de Santiago de Chile
Locations (1):
- Universidad de Santiago de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Scientific background, Objective, Design, and Methods
Supporting Information: Study Protocol, SAP
Time Frame: IPD
URL: https://www.dropbox.com/home/SABE/ActiveStars

DOCUMENTS (1):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03893149/Prot_000.pdf